CLINICAL TRIAL: NCT07272642
Title: A Phase 1, Multicenter Study of the Safety and Imaging of NTH-2403, a Lutetium-177 Radiolabeled Monoclonal Antibody Targeting the LRRC15 Epitope, in Participants With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Phase 1, Multicenter Imaging Study of LNTH-2403 in Participants With Locally Advanced or Metastatic Solid Tumors.
Acronym: DUNP19
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Radiopharm Theranostics, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DUNP19-AU-101
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Imaging; Colorectal Cancer; Head and Neck Squamous Cell Carcinoma; Non-Small Cell Lung Cancer; Triple Negative Breast Cancer (TNBC)
Keywords: imaging; colorectal cancer; Head and Neck squamous cell carcinoma,; non-small cell lung cancer,; triple negative breast cancer
MeSH Terms: conditions — Colorectal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-arm, Single dose, open-label study (Experimental): LNTH-2403 at a dose of 20 mCi(0.74 GBq)
  Interventions: Drug: LNTH-2403

INTERVENTIONS:
Drug: LNTH-2403 — LNTH-2403 (177Lu-DOTA-DUNP19) is a lutetium-177 radiolabeled, fully humanized monoclonal antibody (mAb)

SUMMARY:
LNTH-2403 (177Lu-DOTA-DUNP19) is a lutetium-177 radiolabeled, fully humanized monoclonal antibody (mAb) that binds with high specificity and affinity to leucine-rich repeat containing 15 (LRRC15), a transforming growth factor (TGF) - β-driven biomarker expressed on the cell membrane of cancer cells and/or cancer-associated fibroblasts 9CAFs) in select tumor types. Upon binding, LNTH-2403 is rapidly internalized, such that it can serve as a dual-purpose agent for both non-invasive imaging and radiotheranostic treatment of LRRC15- positive tumors. This first-in-human (FIH) imaging study will evaluate the safety and imaging of LNTH-2403 in participants with locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
This study is a Phase 1, multicenter, open-label, single-dose study of the safety , imaging, and biodistribution of LNTH-2403 in participants with locally advanced or metastatic colorectal cancer (CRC), head and neck squamous cell carcinoma (HNSCC), non-small cell lung cancer (NSLC) (squamous or non-squamous histology), or triple negative breast cancer (TNBC). The study comprises a Screening Period, an Imaging Period, a Safety Follow-up Period, and a Long term Follow-Up Period (LTFU).

The Screening Period will be up to 28 days. Participants will provide written informed consent and eligibility will be confirmed through completion of all screening assessments within 28 days prior to Day 1 administration of LNTH-2403.

The Dosing and Imaging Period encompasses Day 1 through Day 5. Participants will receive a single administration of LNTH-2403 on Day 1. Vital signs, ECGs, and blood sampling will be performed just before LNTH-2403 administration and at the timepoints specified in the protocol after LNTH-2403 administration. Participants will undergo a single whole-body single photon emission computed tomography (SPECT)/CT scan anytime between Days 3 - 5 following administration of LNTH-2403. Blood samples will be collected for LNTH-2403 biodistribution analysis on the day of SPECT/CT imaging.

The Safety Follow-up Period will include a Safety Follow-up Visit, which may be conducted remotely by telephone or telehealth or at the site at the discretion of the Investigator, on Day 28 (±2 days) to assess concomitant medications and EAs/SAEs and to request a post-treatment biopsy sample, if available.

The Long-term Follow-up Period will be conducted to request that participants provide a post-treatment biopsy sample that was obtained ≤ 90 days after LNTH-2403 administration on Day 1and prior to starting a new therapy, if available. The Long-term Follow-up Visit does not need to be completed if a post treatment biopsy sample was obtained at the Safety Follow-up Visit.

Participants are eligible to enroll in another investigational protocol after the SPECT/CT scan and other assessments are performed at the timepoint between Days 3 - 5.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give written informed consent prior to start of any study procedures and assessments and must be willing to comply with all study procedures.
2. Participant is ≥ 18 years of age at the time of signing the informed consent.
3. Participant has a documented history of histopathologically confirmed, locally advanced or metastatic CRC, HNSCC, NSCLC (squamous or non-squamous histology), or TNBC which has progressed despite (or is ineligible for) available standard of care treatment disease
4. Has had a SOC CT or MRI scan within 8 weeks prior to signing informed consent that indicates the presence of at least 1 site of new or residual disease. SOC baseline images must be available for submission to the centralized imaging reader as reference
5. Participant must provide an archived tumor tissue sample.
6. Participant has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
7. Participant has at least 1 visceral lesion that has not been treated with external beam radiation therapy (EBRT).
8. Participants of childbearing potential (CBP) must have a negative beta-human chorionic gonadotropin (β-hCG) test and must not be breastfeeding. Participants of CBP are defined as those who are not surgically sterile or post-menopausal. Participants will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. Participants < 50 years of age who meet the criteria for postmenopausal status without previous surgical sterilization should be considered for further investigation with luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels to confirm serological post-menopausal status.
9. Participants of CBP must agree to use a highly effective method of contraception during the study and for 3 months after the injection of LNTH-2403.
10. Male participants who are able to father a child must agree to avoid impregnating a partner and to adhere to a highly effective method of contraception during the study and for 3 months after the injection of LNTH-2403. All male participants must agree to not donate sperm during the study and for 3 months after the injection of LNTH-2403.

Exclusion Criteria:

1. Has any medical condition that would, in the Investigator's judgment, prevent the participant's full participation in the clinical study due to safety concerns or compliance with clinical study procedures.
2. Has a history of uncontrolled allergic reactions and/or known or expected hypersensitivity to protein therapeutics, LNTH-2403, or any of its excipients.
3. Has inadequate organ functions as reflected in laboratory parameters:

   1. Estimated glomerular filtration rate (eGFR) (calculated using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation) ≤ 50 mL/min/1.73m2
   2. Platelet count <100 x 10^9 /L
   3. Hemoglobin < 9 g/dL
   4. Absolute neutrophil count < 1.0 × 109/L
   5. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3 x upper limit of normal (ULN), or ≥ 5 x ULN for participants with known liver metastases
   6. Total bilirubin ≥ 1.5 x ULN, except for participants with documented Gilbert's syndrome who are eligible if total bilirubin is ≤ 3 x ULN
   7. For participants not taking warfarin or other anticoagulants: international normalized ratio (INR) ≤ 1.5 or prothrombin time (PT) ≤ 1.5 × ULN; and either partial thromboplastin time or activated partial thromboplastin time (PTT or aPTT) ≤ 1.5 × ULN. Participants taking warfarin must be on a stable dose that results in a stable INR < 3.5. Among participants receiving other anticoagulant therapy, PT or aPTT must be within the intended therapeutic range of the anticoagulant.
4. Has clinically significant cardiovascular/ cerebrovascular disease defined as cerebral vascular accident, stroke, carotid artery disease transient ischemic attack (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification Class >II) or serious cardiac arrhythmia.
5. Has a marked baseline prolongation of QT/QTc interval (repeated demonstration of a QTc interval calculated with Fredericia's correction (QTcF) > 470 msec for females and QTcF > 450 msec for males);
6. Has a history of or has additional risk factors for torsade's de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
7. Is participating in an interventional trial or has received an investigational anticancer agent within 5 half-lives of the time of informed consent signature or is expected to enroll in an interventional trial on or before the imaging timepoint during Days 3-5.
8. Has been treated with an LRRC15-targeted investigational product.
9. Has had a PET scan done within 10 physical half-lives of the PET imaging agent prior to receiving study intervention.
10. Is pregnant or breastfeeding.
11. Had or is scheduled to have major surgery within 4 weeks of Day 1 (not including diagnostic laparoscopy).
12. Has a medical history, physical examination, or clinical laboratory test suggestive of a condition, disorder, or disease that could adversely affect drug absorption, distribution, metabolism, or elimination of LNTH-2403, including chronic liver or renal failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of a single dose of LNTH-2403 | 90 days
  Frequency and severity of adverse events (AE)s and serious adverse events (SAEs)using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0

SECONDARY OUTCOMES:
To assess the biodistribution of LNTH-2403 in selected organs and tumor lesions. | 90 days
  Percent of the injected activity per gram of tissue for selected organs and tumor lesions.
  Concentration of LNTH-2403 in blood

OTHER OUTCOMES:
Exploratory: • To explore agreement between LNTH-2403 imaging and LRRC15 and FAP expression by IHC analysis | 90 days
  • The localization of LNTH-2403 on imaging compared with the expression of LRRC15 and FAP in tumor samples as measured by IHC.
Exploratory: To assess the sensitivity, specificity, and accuracy of LNTH-2403 for imaging | 90 days
  The proportion of cases correctly identified by LNTH-2403 as having no metastasis out of the total number of cases confirmed to have no metastasis by SOC imaging methods, such as CT or MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Icon Cancer Centre Hollywood, Nedlands, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No